CLINICAL TRIAL: NCT03367910
Title: Fecal Microbiota Transplantation Using RBX2660 for the Prevention of Recurrent Urinary Tract Infections Due to Multidrug Resistant Organisms
Brief Title: Fecal Microbiota Transplantation (FMT) for MDRO UTI
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); University of Pennsylvania (Other); Duke University (Other); Rush University (Other); Rebiotix Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 201708204
Record Dates: First submitted 2017-12-05; First posted 2017-12-11 (Actual); Results first posted 2022-02-28 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Urinary Tract Infections
Keywords: Urinary tract infection; Multidrug resistant organism; Fecal microbiota transplantation
MeSH Terms: conditions — Urinary Tract Infections | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Intervention Model Description: Participants with eligible MDRO UTIs will receive FMT.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- FMT for MDRO UTI (Experimental): Participants with eligible MDRO UTIs will receive FMT (150mL of RBX2660) via enema.
  Interventions: Drug: Fecal microbiota transplant

INTERVENTIONS:
Drug: Fecal microbiota transplant — 150mL of FMT product RBX2660 delivered via enema
  Other Names: Stool transplant

SUMMARY:
The purpose of this study is to determine the safety and impact of fecal microbiota transplantation (FMT) on the fecal and urine microbiome, urine metabolome, risk of recurrent urinary tract infection (UTI), and persistent multidrug resistant organism (MDRO) colonization of patients with a history of recurrent MDRO UTIs. This is an open label phase 1-2 study.

DETAILED DESCRIPTION:
Multidrug resistant organism (MDRO) infections are increasingly common. The most common type of infection caused by MDROs is urinary tract infections (UTIs). Many MDROs are inhabitants of the colon, and MDROs can contaminate the periurethral area and migrate to the bladder. Patients with MDRO UTI frequently experience multiple relapses and hospitalizations, which both increase the individual's morbidity and mortality and leads to additional MDRO nosocomial spread. There are few options available to prevent MDRO UTIs, and there are limited strategies to identify patients at risk for recurrent MDRO UTI and prevent or reverse MDRO colonization. A potential novel method to reverse MDRO colonization and prevent recurrent UTI would be by repopulating the gut microbiome with "healthy" microbiota by fecal microbiota transplantation (FMT).

In this study, participants with a history of severe, recurrent MDRO UTI will receive FMT. Participants will submit stool and urine specimens pre- and post-FMT, and the effect of FMT on the participants' fecal and urine microbiome, urine metabolome, persistent MDRO colonization, and risk of recurrent UTI will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old.
* Outpatient status at time of FMT.
* History of at least three recurrent UTIs due to an MDRO; at least two recurrent, severe infections due to MDRO requiring hospitalization; or at least two recurrent infections due to MDRO for which only antimicrobials with rate limiting toxicities (see above) are available.
* Be without active infection due to the MDRO at the time of FMT.
* Not be receiving antimicrobials (therapeutic or suppressive) within 48 hours of FMT.

Exclusion Criteria:

* Age <18 years
* Inpatient status at time of FMT
* Ineligible UTI
* >1 organism in urine (other than minimal contaminants)
* Decline to participate
* Recurrent Clostridium difficile infection
* Presence of intra-abdominal devises
* Neutropenia (ANC <500 mm3)
* Intestinal mucosal disruption
* Unlikely to survive 6 months
* Pregnancy or unwillingness to use contraceptives
* Short gut syndrome
* Use of medications that affect intestinal motility
* Gastrointestinal motility disorder
* Inflammatory bowel disease
* Recent abdominal surgery
* Active typhlitis
* Active diverticulitis
* Current gastrointestinal graft versus host disease
* HIV with lack of antiretroviral therapy (ART)
* CD4 count <200 mm3
* Peritoneal dialysis
* Cirrhosis with ascites
* Active intra-abdominal malignancy
* Presence of chronic indwelling foley catheter, chronic suprapubic catheter, or ileal conduit
* Active hepatitis C
* Active hepatitis B
* Presence of ureteral stent
* Active kidney stone that is believed to be a persistent source of bacterial colonization
* Any condition where the investigator feels the risks of FMT outweigh the benefits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2018-02-08 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erik Dubberke, MD, MSPH, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | FMT for MDRO UTI
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | FMT for MDRO UTI
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 1
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Adverse Events During and After FMT
Description: The number, types, severity, and relation of adverse events to study procedures or product will be analyzed.
Time Frame: Six months post-FMT
Measure: Count of Participants; unit: Participants
Arm/Group | FMT for MDRO UTI
Number analyzed (Participants) | 1
Participants | 1

2. Secondary Outcome: Number of Patients With Recurrent UTI Post-FMT
Description: Risk of recurrent UTI post-FMT will be evaluated
Time Frame: Six months post-FMT
Measure: Count of Participants; unit: Participants
Arm/Group | FMT for MDRO UTI
Number analyzed (Participants) | 1
Participants | 1

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | FMT for MDRO UTI
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FMT for MDRO UTI (N=1)
Diarrhea (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-22): https://cdn.clinicaltrials.gov/large-docs/10/NCT03367910/Prot_SAP_000.pdf